CLINICAL TRIAL: NCT03817944
Title: Placebo-controlled Study on Intervention Effect of Coffee on Glucose and Lipid Homeostasis Disorders
Brief Title: Effects of Coffee Consumption on Health Among Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Yu Zhang, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: RCT-Coffee
Record Dates: First submitted 2019-01-23; First posted 2019-01-28 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Health
Keywords: body weight; glucose; lipid; metabolites; gut microbiota
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Warm Water (Placebo Comparator): 300 mL Warm Water per day for 8 weeks
  Interventions: Other: Warm Water
- Caffeinated Coffee (Experimental): 300 mL Caffeinated Coffee per day for 8 weeks
  Interventions: Other: Caffeinated Coffee
- Decaffeinated Coffee (Experimental): 300 mL Decaffeinated Coffee per day for 8 weeks
  Interventions: Other: Decaffeinated Coffee

INTERVENTIONS:
Other: Warm Water — 300 mL Warm Water per day for 8 weeks
  Arms: Warm Water
Other: Caffeinated Coffee — 300 mL Caffeinated Coffee per day for 8 weeks
  Arms: Caffeinated Coffee
Other: Decaffeinated Coffee — 300 mL Decaffeinated Coffee per day for 8 weeks
  Arms: Decaffeinated Coffee

SUMMARY:
The purpose of this study is to research the changes of typical thermal processing food intervention on health outcome, metabolites, and gut microbiota, in order to explore the molecular mechanism of interaction between maillard reaction associated hazards and complex food matrix, and provide scientific basis and reference model for combining food nutrition and safety protection.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, non-occupational exposed healthy volunteers, 18.5<BMI<30 kg/m^2, were screened. If the evaluation of disease history, blood biochemistry and blood routine was normal, the volunteers were considered healthy.

Exclusion Criteria:

* The main exclusion criteria included people with high exposure to cold and fever, recent drug intake (including dietary supplement intake), alcohol intake, vegetarians, pregnancy, high-temperature processed meat and beverages such as coffee and milk tea.

Ages: 17 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 156 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose from baseline | 8 weeks
Change in blood lipids from baseline | 8 weeks

SECONDARY OUTCOMES:
Urinary biomarkers levels of acrylamide, furans, and furfuryl alcohol | 8 weeks; 24 hours
  Urinary levels of environmental pollutants (e.g., acrylamide, furans, and furfuryl alcohol), measured using liquid chromatography-mass spectrometry (LC-MS)
Change of metabolites | 8 weeks
Change in gut microbiota | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang university, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No